CLINICAL TRIAL: NCT04844125
Title: A Multicentric, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of SHR-1209 in Patients With Hypercholesterolemia
Brief Title: SHR - 1209 Treatment Efficacy and Safety of the Patients With Hypercholesterolemia Ⅲ Period Clinical Research
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1209-303
Record Dates: First submitted 2021-04-02; First posted 2021-04-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-05

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Background Lipolowering therapy in combination with SHR-1209/ placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1209 (Experimental)
  Interventions: Drug: SHR-1209
- SHR-1209 Placebo (Placebo Comparator)
  Interventions: Drug: SHR-1209 Placebo

INTERVENTIONS:
Drug: SHR-1209 — SHR-1209
  Arms: SHR-1209
Drug: SHR-1209 Placebo — SHR-1209 Placebo
  Arms: SHR-1209 Placebo

SUMMARY:
This study is ongoing to evaluate the efficacy and safety of SHR-1209 in patients with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

1. Any male or female aged between 18 and 80 on the date of signing the informed consent;
2. Diagnosed as hypercholesterolemia ;
3. Fasting triglyceride was less than 5.6 mmol/L during screening:
4. Understand the study procedures and methods, volunteer to participate in the study, and sign the informed consent.

Exclusion Criteria:

1. A history of the following diseases or treatments during the screening period:

   1. Known allergies to PCSK9 inhibitors or test drugs, or severe allergic reactions to other antibody drugs in the past;
   2. Participated in clinical studies of other drug interventions within the last 1 month (except for patients who failed in screening), or those who are within 5 half-lives of the drug before screening (whichever is longer);
2. Any of the laboratory test indicators meets the following criteria:

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) was more than 3 times the upper limit of normal value (ULN), and total bilirubin was more than 2 times ULN during the screening period or at random;
   2. The creatine kinase (CK) was more than 3 times of ULN during the screening period or at random;
3. Have used the following drugs:

   1. PCSK9 inhibitors had been used in the previous 6 months;
   2. Continuous systemic corticosteroid therapy with doses exceeding or equivalent to 10mg of prednisone (oral or intravenous) within the previous 3 months was screened.
4. Other circumstances:

   1. Women of reproductive age who are fertile but did not use contraception within 4 weeks before the screening period;Women who are pregnant or breastfeeding;Not agreed during the trial or at 24 weeks after the last dose
   2. Subjects who are considered by the investigator to have any unsuitable factors for participating in the study or who have poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
12 weeks Percentage change in serum LDL-C levels from baseline. | 12 weeks

SECONDARY OUTCOMES:
12 weeks Absolute Changes in serum LDL-C levels from baseline； | 12 weeks
12 weeks Percentage change of non-HDL-C relative to baseline； | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangzhou, China

REFERENCES:
- [Derived] Li L, Zhou Y, Deng C, Sheng J, Peng D, Ling Z, Wang L, Dai C, Huang K, Lian Q, Yu Z, Yang H, Hu Y, Dong Y, Wang N, Wang Z, Zhang W, Han X, Yao Z, Liu Q, Liang Y, Xu B, Wang Y, Zhong T, Chen J. Recaticimab in adult heterozygous familial hypercholesterolaemia (REMAIN-3): a multicentre, randomized, double-blind, placebo-controlled Phase 3 study. Cardiovasc Res. 2025 Oct 24;121(12):1856-1864. doi: 10.1093/cvr/cvaf155. PMID 40911402
- [Derived] Shu C, Wang Y, Feng S, Yang S, Shen K. Population Pharmacokinetics and Pharmacodynamics Modeling for the Use of Recaticimab in Healthy Volunteers and Patients with Hypercholesterolemia. Clin Pharmacokinet. 2025 Sep;64(9):1341-1355. doi: 10.1007/s40262-025-01512-5. Epub 2025 Jun 30. PMID 40587053